CLINICAL TRIAL: NCT04235439
Title: A Glucose Clamp Trial Investigating the Biosimilarity of Gan & Lee Insulin Lispro Injection With Both EU - Approved and US - Licensed Humalog® in Healthy Male Subjects
Brief Title: PK/PD Biosimilarity Study of Gan & Lee Insulin Lispro Injection vs. EU and US Humalog® in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GL - LSP - 1006
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Insulin; Lispro; Diabetes Mellitus; Basal; Bolus
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — gallium nitrate

STUDY DESIGN:
Intervention Model Description: This is a phase 1 trial. The trial is a single center, randomized, doubleblind, single dose, there treatment, three period crossover, 12 - hour euglycaemic glucose clamp trial in healthy male subjects.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gan & Lee Insulin Lispro Injection (Experimental): Insulin lispro, 3 mL cartridge in prefilled pen, 100 units/mL (U-100)
  Interventions: Drug: Gan & Lee Insulin Lispro Injection
- EU - approved Humalog ® (Active Comparator): Insulin lispro (product approved and marketed in the EU), 3 mL cartridge in prefilled Kwikpen®, 100 units/mL (U-100)
  Interventions: Drug: Gan & Lee Insulin Lispro Injection
- US - licensed Humalog ® (Active Comparator): Insulin lispro (product approved and marketed in the US), 3 mL cartridge in prefilled Kwikpen®, 100 units/mL (U-100)
  Interventions: Drug: Gan & Lee Insulin Lispro Injection

INTERVENTIONS:
Drug: Gan & Lee Insulin Lispro Injection — All three IMPs will be administered as a 0.2 U/kg single dose subcutaneously in the periumbilical area by use of a disposable prefilled pen.
  Other Names: EU - approved Humalog ®; US - licensed Humalog ®

SUMMARY:
Primary objective:

To demonstrate pharmacokinetic (PK) and pharmacodynamic (PD) equivalence of Gan & Lee Insulin Lispro Injection with both EU - approved Humalog® and US - licensed Humalog® (Reference Products) in healthy male subjects

Secondary objectives:

To compare the PK and PD parameters of the three insulin lispro preparations

To evaluate the single dose safety and local tolerability of the three insulin lispro preparations

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial related activities. Trial related activities are any procedures that would not have been done during normal management of the subject
2. Healthy male subjects
3. Age between 18 and 64 years, both inclusive
4. Body Mass Index (BMI) between 18.5 and 29.0 kg/m^2, both inclusive
5. Fasting plasma glucose concentration <= 5.5 mmol/L (100 mg/dL) at screening
6. Considered generally healthy upon completion of medical history and screening safety assessments, as judged by the Investigator

Exclusion Criteria:

1. Known or suspected hypersensitivity to IMP(s) or related product
2. Previous participation in this trial. Participation is defined as randomized
3. Receipt of any medicinal product in clinical development within 30 days before randomization in this trial
4. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
5. Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the Investigator
6. Any history or presence of clinically relevant comorbidity, as judged by the Investigator
7. Signs of acute illness as judged by the Investigator
8. Any serious systemic infectious disease during four weeks prior to first dosing of the trial drug, as judged by the Investigator
9. Clinically significant abnormal screening laboratory tests, as judged by the Investigator
10. Elevation of serum ALT> 10% above the ULN, or elevation of serum AST or serum bilirubin >20% above the ULN. (Note: Elevation of bilirubin is considered acceptable in case of Gilbert's disease and should be evaluated in clinical context)
11. Elevation of serum creatinine > ULN, or elevation of serum urea > 10% above ULN
12. Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or > 89 mmHg (one repeat test will be acceptable in case of suspected white-coat hypertension)
13. Symptoms of arterial hypotension
14. Heart rate at rest outside the range of 50-90 beats per minute
15. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator
16. Increased risk of thrombosis, e.g. subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator
17. Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 24 grams alcohol/day (on average)
18. A positive result in the alcohol and/or urine drug screen at the screening visit
19. Smoking more than 5 cigarettes or the equivalent per day
20. Inability or unwillingness to refrain from smoking and use of nicotine substitute products one day before and during the inpatient period
21. Positive test for Hepatitis Bs antigen
22. Positive test for Hepatitis C antibodies. (Presence of Hepatitis C antibodies will not lead to exclusion if liver function tests are normal and a hepatitis C polymerase chain reaction is negative)
23. Positive result to the test for HIV-1/2 antibodies or HIV-1 antigen
24. Any medication (prescription and non-prescription drugs) within 7 days before IMP administration and/or anticoagulant therapy
25. Blood donation or blood loss of more than 500mL within the last 3 months
26. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation

Explanatory note on Exclusion Criterion 24: With the exception of paracetamol or NSAIDs for occasional use to treat acute pain, as judged by the Investigator.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
AUCins.0-12h | 0 to 12 hours
  PK Endpoint: The area under the insulin concentration curve from 0 to 12 hours.
Cins.max | 0 to 12 hours
  PK Endpoint: The maximum observed insulin concentration.
AUCGIR.0-12h | 0 to 12 hours
  PD endpoint: The area under the glucose infusion rate curve from 0 to 12 hours.
GIRmax | 0 to 12 hours
  PD endpoint: The maximum glucose infusion rate.

SECONDARY OUTCOMES:
AUCins.0-2h | 0 to 2 hours
  PK endpoint: The area under the insulin concentration curve from 0 to 2 hours
AUCins.0-4h | 0 to 4 hours
  PK endpoint: The area under the insulin concentration curve from 0 to 4 hours
AUCins.0-6h | 0 to 6 hours
  PK endpoint: The area under the insulin concentration curve from 0 to 6 hours
AUCins.6-12h | 6 to 12 hours
  PK endpoint: The area under the insulin concentration curve from 0 to 12 hours
AUCins.0-∞ | 0 to 12 hours
  PK endpoint: The area under the insulin concentration-time curve from 0 hours to infinity
tins.max | 0 to 12 hours
  PK endpoint: The time to maximum observed insulin concentration t½, terminal serum elimination half-life calculated as t½=ln2/λz
t50%-ins(early) | 0 to 12 hours
  PK endpoint: The time to half-maximum insulin concentration before Cins.max
t50%-ins(late) | 0 to 12 hours
  PK endpoint: The time to half-maximum insulin concentration after Cins.max
t½ | 0 to 12 hours
  PK endpoint: The terminal serum elimination half-life calculated as t½=ln2/λz
λz | 0 to 12 hours
  PK endpoint: The terminal elimination rate constant of insulin
AUCGIR.0-2h | 0 to 2 hours
  PD endpoint: The area under the glucose infusion rate curve from 0 to 2 hours
AUCGIR.0-4h | 0 to 4 hours
  PD endpoint: The area under the glucose infusion rate curve from 0 to 4 hours
AUCGIR.0-6h | 0 to 6 hours
  PD endpoint: The area under the glucose infusion rate curve from 0 to 6 hours
AUCGIR.6-12h | 6 to 12 hours
  PD endpoint: The area under the glucose infusion rate curve from 6 to 12 hours
tGIR.max | 0 to 12 hours
  PD endpoint: The time to maximum glucose infusion rate
tGIR.50%-early | 0 to 12 hours
  PD endpoint: The time to half-maximum glucose infusion rate before GIRmax
tGIR.50%-late | 0 to 12 hours
  PD endpoint: The time to half-maximum glucose infusion rate after GIRmax
PD endpoint | 0 to 12 hours
  time to onset of action
Safety and Local Tolerability | 0 to 12 hours
  Number of participants experiencing treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jia Lu, PhD, Study Director — Gan & Lee Pharmaceuticals, USA; Leona Plum - Mörschel, Dr. med, Principal Investigator — Profil Mainz GmbH & Co KG
Locations (1):
- Profil Mainz GmbH & Co. KG, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen W, Lu J, Plum-Morschel L, Andersen G, Zijlstra E, He A, Xie T, Li L, Hao C, Gan Z, Heise T. Pharmacokinetic and pharmacodynamic bioequivalence of Gan & Lee insulin analogues aspart (rapilin(R)), lispro (prandilin(R)) and glargine (basalin(R)) with EU- und US-sourced reference insulins. Diabetes Obes Metab. 2023 Dec;25(12):3817-3825. doi: 10.1111/dom.15281. Epub 2023 Sep 21. PMID 37735841